CLINICAL TRIAL: NCT01083199
Title: Global Performance Evaluation of the AMS CONTINUUM™ Device in Facilitating Vesico-Urethral Anastomosis Following a Radical Prostatectomy
Brief Title: Global Performance Evaluation of the AMS CONTINUUM™ Device
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: American Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PE0702
Record Dates: First submitted 2010-03-04; First posted 2010-03-09 (Estimated); Results first posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2011-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Radical Prostatectomy; Vesico-Urethral Anastomosis
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Continuity of Patient Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CONTINUUMTM (Experimental)
  Interventions: Device: CONTINUUM™

INTERVENTIONS:
Device: CONTINUUM™ — Performance of CONTINUUM™ in facilitating the vesico-urethral anastomosis following radical prostatectomy.
  Other Names: Anastomosis Device

SUMMARY:
1. To evaluate Device performance in providing mucosa to mucosa apposition to facilitate sustainable vesico-urethral anastomosis during a radical prostatectomy procedure.
2. To assess clinical outcomes of the Device in facilitating the vesico-urethral anastomosis following a radical prostatectomy.

DETAILED DESCRIPTION:
Radical prostatectomy (RP) is the most utilized surgical treatment option for localized prostate cancer due to the multi-focal nature of the disease. RP is most suitable for otherwise healthy men whose cancer is limited to a small area. The RP procedure involves removing the prostate gland, seminal vesicles and nearby lymph nodes. One of the most technically challenging and critical aspects in all of these surgical approaches is reconstruction of the interrupted urinary tract by hand sewing the vesico-urethral anastomosis. This is where the bladder neck is sewn to the urethra after the prostate has been removed.

CONTINUUM™ (study Device) is to be used as part of the RP procedure by facilitating the approximation of the bladder neck and urethral stump. The Device brings together and holds the tissue in place until adequate natural healing of the vesico-urethral anastomosis occurs thereby minimizing extravasation. The Device also provides a conduit for drainage of urine from the bladder out the urethra during tissue healing.

The concept of the CONTINUUM™ device and the feasibility of its operation have been successfully tested in animal and human studies. Pilot clinical studies in the United States (G060095) found that the majority of subjects who received and were discharged with the Device demonstrated a water-tight vesico-urethral anastomosis at the first Device removal visit. Additionally, no unanticipated adverse device effects (UADEs) were reported. The focus of the proposed study is to further verify the performance of the Device in global research centers.

ELIGIBILITY:
Inclusion Criteria:

* All males ≥ 40 years old who are indicated for a radical prostatectomy will be eligible to participate in the study

Exclusion Criteria:

* If contraindicated for surgery
* Inability to understand the study or a history of non-compliance with medical advice
* Unwilling or unable to sign an Informed Consent Form (ICF)
* A history of:

  1. Recurrent urinary tract infections (UTI)
  2. Recurrent stricture disease
* Neurological disease with a history of bladder dysfunction (e.g., Parkinson's disease)
* Uncontrolled insulin-dependent diabetes
* Chemotherapy within the past 6 months
* Non-topical steroid use within the past 6 months
* Allergy to nitinol, nickel, titanium or silicone

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-10; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Liatsikos, MD, Principal Investigator — University of Patras; Carlos Hernandez, MD, Principal Investigator — Hospital University Gregorio Maranon
Locations (2):
- University of Patras, Rio-Patras, Greece
- Hospital University Gregorio Maranon, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AMS CONTINUUM™ Device
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AMS CONTINUUM™ Device
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.7 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10

OUTCOME MEASURES:

1. Primary Outcome: Successful Device Placement
Description: Successful Device placement was defined as the establishment of a water-tight anastomosis immediately post-Device placement.
Time Frame: During Radical Prostatectomy
Measure: Number; unit: participants
Arm/Group | Continuum Device
Number analyzed (Participants) | 10
participants | 10

2. Primary Outcome: Functionally Adequate Vesico-urethral Anastomosis Within 21 Days Post-procedure in Subjects With Successful Device Placement
Description: Device removal was first attempted at the 7-day window; if extravasation was noted, the subject returned for a second attempt at the 14-day window. If extravasation was noted at the first and second attempts, the subject could then return for a 3rd and final removal at the 21-day window.
  The following defines the timeframe of each removal attempt:
  * 7-day window (7-10 days post-implant)
  * 14-day window (13-15 days post-implant)
  * 21-day window (19-21 days post-implant)
Time Frame: 7-21 days post-Device placement
Measure: Number; unit: participants with device removal by 21d
Arm/Group | AMS CONTINUUM™ Device
Number analyzed (Participants) | 10
participants with device removal by 21d | 10

3. Secondary Outcome: Intraoperative/Postoperative Parameters
Time Frame: At Device placement
Reporting Status: Not Posted

4. Secondary Outcome: Percentage of Subjects Demonstrating Functionally Adequate Anastomosis at the 1st and 2nd Device Removal Visits
Time Frame: 7 and 14 days post-Device placement
Reporting Status: Not Posted

5. Secondary Outcome: Incontinence Rate and I-QOL Score
Time Frame: Baseline, 6-week, 6 and 12-month evaluations
Reporting Status: Not Posted

6. Secondary Outcome: Bladder Neck Contracture (BNC) Rate
Time Frame: Subjects that develop BNC between the scheduled follow-up visits at 6 weeks, 6 and 12 months post-device removal
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | AMS CONTINUUM™ Device
Serious Adverse Events (participants affected / at risk) | 6/10
Other Adverse Events (participants affected / at risk) | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMS CONTINUUM™ Device (N=10)
Hemorrhage (Vascular disorders) | 1 (1)
Migration (Renal and urinary disorders) | 1 (1)
Separation/Distruption of Anastomosis (Renal and urinary disorders) | 4 (4)
Urinary Retention (Renal and urinary disorders) | 1 (1)
Urinary Tract Infection (UTI) (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AMS CONTINUUM™ Device (N=10)
False Passage (Renal and urinary disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 5 (6)
Rectal Injury (Renal and urinary disorders) | 1 (1)
Separation/Disruption of Anastomosis (Renal and urinary disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No